CLINICAL TRIAL: NCT04196322
Title: Hyperglycemia as a Prognostic Factor In Acute Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: El Zaitoun Specialized Hospita
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Acute Ischemic Stroke Patients
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controlled
  Interventions: Other: observational study
- Uncontrolled
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Background: Hyperglycemia is encountered in 20% to 40% of acute stroke patients, with or without a pre-morbid diagnosis of diabetes mellitus. Hyperglycemia is a risk factor for infarct expansion and poor outcome through the first 72 hours of onset in both diabetics and non-diabetics patients. This study was done to evaluate the glycemic status after acute ischemic stroke and assess its rule in influencing stroke outcome as regards the duration of hospital stay, motor deficit and mortality.

Methods: This retrospective study was conducted in Elzaiton specialized hospital from June 2016 to June 2017on 80 patients after approval of local medical ethical committee. Patients with acute ischemic stroke without other major comorbidities within 24 hours of onset of symptoms were included and divided into two groups, controlled group (Random blood suger not more than 150 mg/dl) and uncontrolled group ( Random blood suger more than 150 mg/dl). All patients were evaluated for GCS as a primary outcome and for hemorrhagic transformation, hospital stay duration, mechanical ventilation, need for vasopressors,hospital stay and mortality as secondary outcomes.

DETAILED DESCRIPTION:
Patients and Methods This study was prospective study conducted in Elzaiton specialized hospital and Ain Shams University from june2016 to June 2017on 80 patients after approval of local medical ethical committee

All patients was subjected to the following

1. Full clinical history …age, sex, weight and medical history
2. GCS and motor deficit
3. Random blood glucose level at admission and 4-6 times daily during hospital stay
4. HbA1c on admission
5. Hemodynamic monitoring
6. Duration of hospital stay
7. Thirty day mortality
8. Other laboratory investigation to rule out other similar cause
9. Follow up hemorrhagic transformation Study tools: Patients with acute ischemic stroke without other major comorbidities within 24 hours of onset of symptoms will be evaluated.

On ICU admission the random blood sugar was recorded and categorized to less than 150mg/dl (accepted) and more than 150mg/dl(not controlled). Also serial Random blood sugar daily was recorded and categorized to accepted or good control if less than 150mg/dl and not controlled if more than 150mg/dl.

Patients were divided into 2 groups Patients with accepted random blood sugar at admission and controlled blood sugar during hospital stay.

Patients with increased random blood sugar at admission and poor blood sugar control during hospital stay.

These data were collected and patients were observed as regards duration of hospital stay,hemorrhagic transformation, hospital stay duration and 30-days mortality

ELIGIBILITY:
Inclusion criteria

* Age: 40-70years
* Sex: Any sex
* Patients with acute ischemic stroke without other major comorbidities within 24 hours of onset of symptoms were evaluated.

Exclusion criteria

* Subdural heamatoma, metabolic causes or transient ischemic attack
* Sub arachnoid heamorrage
* Heamorragic stroke
* Patients with major comorbidities at admission as end stage liver disease, end stage renal disease and malignant hypertension
* Patients with hyperglycemia at admission and controlled blood sugar during hospital stay
* Patients with DKA or hypoglycemia (RBS less than 70 mg dl)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke without other major comorbidities within 24 hours of onset of symptoms will be evaluated.
  At ICU admission the random blood sugar was recorded and categorized to less than 150mg/dl (accepted) and more than 150mg/dl(not controlled). Also serial Random blood sugar daily was recorded and categorized to accepted or good control if less than 150mg/dl and not controlled if more than 150mg/dl.
  Patients were divided into 2 groups Patients with accepted random blood sugar at admission and controlled blood sugar during hospital stay (B) Patients with increased random blood sugar at admission and poor blood sugar control during hospital stay These data were collected and patients were observed as regards duration of hospital stay, motor deficit improvement or worsening using Rating scale for muscle strength
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
GCS | 30 days
  GCS was assessed for 30 days

SECONDARY OUTCOMES:
30 days mortality | 30 days
  30 days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No